CLINICAL TRIAL: NCT02458456
Title: Isometric Handgrip Exercise for Blood Pressure Management. A Randomized, Controlled Trial
Brief Title: Isometric Handgrip Exercise for Blood Pressure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England, Australia (Other)
Responsible Party: Principal Investigator, Deb Carlson, Sponsor-Investigator, University of New England
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UNewEngland1
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- IHG 5% Hypertensive (Sham Comparator): Participants who are either un-medicated pre-hypertensive or medicated for blood pressure management conducting isometric resistance training using a hand dynamometer at 5% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training
- IHG 30% Hypertensive (Experimental): Participants who are either un-medicated pre-hypertensive or medicated for blood pressure management conducting isometric resistance training using a hand dynamometer at 30% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training
- IHG 30% Normotensive (Experimental): Participants who are normotensive conducting isometric resistance training using a hand dynamometer at 30% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training
- IHG 5% Normotensive (Sham Comparator): Participants who are normotensive conducting isometric resistance training using a hand dynamometer at 5% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training
- IHG 10% Hypertensive (Experimental): Participants who are either un-medicated pre-hypertensive or medicated for blood pressure management conducting isometric resistance training using a hand dynamometer at 10% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training
- IHG 10% Normotensive (Experimental): Participants who are normotensive conducting isometric resistance training using a hand dynamometer at 10% of their maximum voluntary contraction. Participants with perform 4 x 2 minutes isometric handgrip exercises 3 times per week under supervision for 8 weeks.
  Interventions: Other: Isometric resistance training

INTERVENTIONS:
Other: Isometric resistance training — Isometric exercise using a hand dynamometer.

SUMMARY:
The aim of this project is to conduct a randomised controlled trial to assess the effect of performing isometric exercise using a handgrip dynamometer on blood pressure.

DETAILED DESCRIPTION:
Recent meta-analyses suggest isometric resistance training (IRT) may be superior to aerobic exercise for lowering blood pressure. A randomised controlled study will be conducted with participants who are either pre-hypertensive, blood pressure between 120/80 and 140/90, or on medication to control their blood pressure. Previous studies have utilised a sedentary control so we intend to use a sham group to determine if it can be used as a working control for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Those within the required age limits, both normotensive, pre-hypertensive, and those medicated for blood pressure management.

Exclusion Criteria:

* Younger than 30 years and older than 70 years; those deemed not to have the capacity to voluntarily participate, unable to participate under their doctor's recommendation, or with arthritis or carpal tunnel syndrome who may aggravate their condition with handgrip exercise.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Baseline and 8 weeks

SECONDARY OUTCOMES:
Compare and contrast changes in blood pressure between the 5% maximum voluntary contraction (MVC) and 30% MVC hypertensive groups | Baseline and 8 weeks
Compare and contrast blood pressure changes between the 30% maximum voluntary contraction (MVC) hypertensive and 30% MVC normotensive groups | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Smart, PhD, Principal Investigator — University of New England
Locations (1):
- University of New England, Armidale, New South Wales, Australia

REFERENCES:
- [Background] Carlson DJ, Dieberg G, Hess NC, Millar PJ, Smart NA. Isometric exercise training for blood pressure management: a systematic review and meta-analysis. Mayo Clin Proc. 2014 Mar;89(3):327-34. doi: 10.1016/j.mayocp.2013.10.030. PMID 24582191